CLINICAL TRIAL: NCT01811303
Title: Effects of Added D-fagomine on Glycaemic Responses to Sucrose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioglane (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RSSL SSID P12-06545
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Reduction of Post-prandial Glycaemic Response
MeSH Terms: interventions — fagomine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-fagomine (Experimental): Measure the changes produced on the postprandial Glycaemic response to 50 g of sucrose containing 40 mg D-fagomine, in 200 ml water
  Interventions: Other: D-fagomine
- Control (Placebo Comparator): Sucrose 50 g without d-fagomine, in 200 ml water
  Interventions: Other: D-fagomine

INTERVENTIONS:
Other: D-fagomine — Measure the changes produced on the postprandial Glycaemic response

SUMMARY:
The purpose of this study is to determine whether D-fagomine affects glycaemic responses to sucrose (commercial white sugar)and quantify the response

DETAILED DESCRIPTION:
This is a two treatment randomized double-blind crossover study, with each test product replicated twice.

Randomization: Subjects will be randomized to a Williams Latin square design balanced for treatment order.

Washout: 2 days or more (may return on day 3)

Run-in: High carbohydrate diet guidance (>150 g/d) 1 day before treatment, recommend same sized dinner the previous night (no food record collection required)

Drop-outs: Subjects who have dropped out before visit 2 will be replaced by another subject randomized in their place (the new subject will complete all treatments)

Subjects will report after an overnight (12 hour) fast for baseline sample collection, and will consume the test product in a fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (not less than 40% Male)
* Aged 18 - 55 years
* Have a body mass index between 18.5 to 29.99 kg/m2
* Healthy, non-diabetic, no gastric bypass surgery
* Have a fasting plasma glucose (finger-stick) <100 mg/dl (<5.5 mmol/L)
* Willing and able to provide written informed consent

Exclusion Criteria:

* Smokers
* Allergic to dairy or soy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rungano Munyuki, Principal Investigator — Reading Scientific Services Ltd.
Locations (1):
- Reading Scientific Services Ltd., Reading, United Kingdom

REFERENCES:
- [Background] Gomez L, Molinar-Toribio E, Calvo-Torras MA, Adelantado C, Juan ME, Planas JM, Canas X, Lozano C, Pumarola S, Clapes P, Torres JL. D-Fagomine lowers postprandial blood glucose and modulates bacterial adhesion. Br J Nutr. 2012 Jun;107(12):1739-46. doi: 10.1017/S0007114511005009. Epub 2011 Oct 3. PMID 22017795
- [Background] Amezqueta S, Galan E, Vila-Fernandez I, Pumarola S, Carrascal M, Abian J, Ribas-Barba L, Serra-Majem L, Torres JL. The presence of D-fagomine in the human diet from buckwheat-based foodstuffs. Food Chem. 2013 Feb 15;136(3-4):1316-21. doi: 10.1016/j.foodchem.2012.09.038. Epub 2012 Sep 18. PMID 23194529

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of adults volunteers done by RSSL, in Reading (United Kingdom), under GCP.
Pre-assignment Details: There was 15 subjects screened that all were complying with the eligibility criteria. Finally only 14 subjects were involved in the study and analysed as far the study was planned to involve 12 subjects. All 14 subjects received the treatment randomized to a William's Latin square design balanced for treatment order.
Groups:
- Placebo, Placebo, Treatment, Treatment: The subjects receive placebo in the first two interventions.
- Treatment, Treatment, Placebo, Placebo: The subjects receive treatment in the first two interventions
- Placebo, Treatment, Placebo, Treatment: The subjects receive placebo or treatment in each intervention alternatively, starting with placebo.
- Treatment, Placebo, Treatment, Placebo: The subjects receive placebo or treatment in each intervention alternatively, starting with treatment.
Period: First Intervention (1 Day)
Arm/Group | Placebo, Placebo, Treatment, Treatment | Treatment, Treatment, Placebo, Placebo | Placebo, Treatment, Placebo, Treatment | Treatment, Placebo, Treatment, Placebo
Started | 4 | 4 | 4 | 2
Completed | 4 | 4 | 4 | 2
Not Completed | 0 | 0 | 0 | 0
Period: Washout (2 Days or More)
Arm/Group | Placebo, Placebo, Treatment, Treatment | Treatment, Treatment, Placebo, Placebo | Placebo, Treatment, Placebo, Treatment | Treatment, Placebo, Treatment, Placebo
Started | 4 | 4 | 4 | 2
Completed | 4 | 4 | 4 | 2
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Placebo, Placebo, Treatment, Treatment | Treatment, Treatment, Placebo, Placebo | Placebo, Treatment, Placebo, Treatment | Treatment, Placebo, Treatment, Placebo
Started | 4 | 4 | 4 | 2
Completed | 4 | 4 | 4 | 2
Not Completed | 0 | 0 | 0 | 0
Period: Washout (2 Days or More)
Arm/Group | Placebo, Placebo, Treatment, Treatment | Treatment, Treatment, Placebo, Placebo | Placebo, Treatment, Placebo, Treatment | Treatment, Placebo, Treatment, Placebo
Started | 4 | 4 | 4 | 2
Completed | 4 | 4 | 4 | 2
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | Placebo, Placebo, Treatment, Treatment | Treatment, Treatment, Placebo, Placebo | Placebo, Treatment, Placebo, Treatment | Treatment, Placebo, Treatment, Placebo
Started | 4 | 4 | 4 | 2
Completed | 4 | 4 | 4 | 2
Not Completed | 0 | 0 | 0 | 0
Period: Washout (2 Days or More)
Arm/Group | Placebo, Placebo, Treatment, Treatment | Treatment, Treatment, Placebo, Placebo | Placebo, Treatment, Placebo, Treatment | Treatment, Placebo, Treatment, Placebo
Started | 4 | 4 | 4 | 2
Completed | 4 | 4 | 4 | 2
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention (1 Day)
Arm/Group | Placebo, Placebo, Treatment, Treatment | Treatment, Treatment, Placebo, Placebo | Placebo, Treatment, Placebo, Treatment | Treatment, Placebo, Treatment, Placebo
Started | 4 | 4 | 4 | 2
Completed | 4 | 4 | 4 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- D-fagomine (All Study Participants): Measure the changes produced on the postprandial Glycaemic response to 50 g of sucrose containing 40 mg D-fagomine, in 200 ml water vs placebo.
Arm/Group | D-fagomine (All Study Participants)
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Glycaemic Response Index
Description: On each intervention, the volunteer measured a baseline fasting blood sugar measurement for that day and repeated this approximately 5 minutes later so that two fasting measurements were obtained under the supervision of staff. All of the subsequent measurements were assessed against the average of the two baseline readings. Each subject was then presented with a test product and they were instructed to consume the whole amount within a fifteen-minute period. Each volunteer then took a blood sugar readings at 15, 30, 45, 60, 90 and 120 minutes following the initiation of consumption of the test product. Measurements were taken using the Ascensia Contour, Blood Glucose Monitoring Systems (Bayer), which analysed the blood sample and provided a blood glucose reading in mmol/l. The AUC is calculated using the trapezoid rule and the final outcome is the incremental area under the curve for the arm expressed as a percent of the average response for the control by the same subject.
Time Frame: 120 minutes
Population: The number of participants >10, the repetitions >= 2 and also other variables was determined based on F. Brouns et al., Glycaemic index methodology,Nutrition Research Reviews (2005), 18, 145-171. Also was considered the advice and previous GI studies from RSSL based on master protocol GIMST09.
Measure: Mean (95% Confidence Interval); unit: percentage of AUC fagomine/AUC control
Groups:
- Change D-fagomine/Control AUC at 60 Min: Determine the relative change in the Glycaemic response between sucrose with D-fagomine and sucrose without D-fagomine in the first 60 minutes (postprandial). Calculated on incremental Area Under the Curve (AUC) from the individual glucose measurements in capillary blood, and evaluated by repeated measures ANOVA.
- Change D-fagomine/Control AUC at 120 Min: Determine the relative change in the Glycaemic response between sucrose with D-fagomine and sucrose without D-fagomine in the first 120 minutes (postprandial). Calculated on incremental Area Under the Curve (AUC) from the individual glucose measurements in capillary blood, and evaluated by repeated measures ANOVA.
Arm/Group | Change D-fagomine/Control AUC at 60 Min | Change D-fagomine/Control AUC at 120 Min
Number analyzed (Participants) | 14 | 14
percentage of AUC fagomine/AUC control | 73.28 [63.66 to 82.90] | 83.45 [67.73 to 99.17]
Statistical Analysis 1: Comparison: Change D-fagomine/Control AUC at 60 Min; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: Change D-fagomine/Control AUC at 120 Min; Test type: Superiority or Other; p < 0.016, ANOVA

2. Secondary Outcome: Maximum Blood Glucose Concentration (C Max) Over the Baseline
Description: Determine the glucose C max of Sucrose with D-fagomine over the baseline.
  The blood glucose maximum concentration (C-Max) expressed in mmol/L of the average response for a 50g sucrose, over the baseline.
  Calculation of the outcome is= (Measure glucose C-Max - Measure glucose baseline)
Time Frame: Usually in the range of 30-45 minutes
Measure: Mean (Standard Error); unit: mmol/L
Groups:
- D-fagomine: Determination of glucose Cmax over the Baseline of the treatment: sucrose 50 g + 200 ml water + 40 mg D-fagomine. Blood glucose concentration expressed in mmol/l.
- Control: Determination of glucose Cmax over the Baseline of the control: sucrose 50 g + 200 ml water. Blood glucose concentration expressed in mmol/l.
Arm/Group | D-fagomine | Control
Number analyzed (Participants) | 14 | 14
mmol/L | 2.3 (0.19) | 3.6 (0.37)

ADVERSE EVENTS:
Groups:
- D-fagomine (All Study Participants): Measure the changes produced on the postprandial Glycaemic response to 50 g of sucrose containing 40 mg D-fagomine, in 200 ml water.
- Placebo - Control (All Study Participants): Measure the changes produced on the postprandial Glycaemic response to 50 g sucrose in 200 ml water (without d-fagomine)
Arm/Group | D-fagomine (All Study Participants) | Placebo - Control (All Study Participants)
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No